CLINICAL TRIAL: NCT06173765
Title: Understanding Dose Related Effects of Strawberry Intake on Chronic Inflammation, Oxidative Stress, and Their Relationship With Endothelial Function and Insulin Sensitivity
Brief Title: Understanding Dose Related Effects of Strawberry
Acronym: STRW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Principal Investigator, Britt Marie Burton-Freeman, Principal Investigator, Clinical Nutrition Research Center, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2021-98
Record Dates: First submitted 2023-05-22; First posted 2023-12-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Pre-diabetes; Insulin Sensitivity; Insulin Resistance; Inflammation
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Inflammation | interventions — Powders

STUDY DESIGN:
Intervention Model Description: a 3 arm, randomized, controlled parallel design using the control arm from the USDA parallel study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 36g of strawberry (Experimental): High dose intervention
  Interventions: Other: freeze-dried whole strawberry powder 36 g powder
- 12g of strawberry (Experimental): Low dose intervention
  Interventions: Other: freeze-dried whole strawberry powder 12 g
- 0g of strawberry (Placebo Comparator): Control
  Interventions: Other: freeze-dried control powder 0 g strawberry

INTERVENTIONS:
Other: freeze-dried whole strawberry powder 36 g powder — After day 1 measurements, subjects will be given their first intervention drink (powder plus water) according to their randomization to 3 cup FW equivalent of strawberries. The freeze-dried whole strawberry powder (36 g powder) requested from the California Strawberry Commission.
  All drinks will be standardized to 41 g powder to match USDA Control arm.
  Arms: 36g of strawberry
Other: freeze-dried whole strawberry powder 12 g — After day 1 measurements, subjects will be given their first intervention drink (powder plus water) according to their randomization to 1 cup FW equivalent of strawberries. The freeze-dried whole strawberry powder (12 g powder) requested from the California Strawberry Commission.
  All drinks will be standardized to 41 g powder to match USDA Control arm.
  Arms: 12g of strawberry
Other: freeze-dried control powder 0 g strawberry — After day 1 measurements, subjects will be given their first intervention drink (powder plus water) according to their randomization to 0 cup FW equivalent of strawberries. The freeze-dried powder is used as a control.
  All drinks will be standardized to 41 g powder to match USDA Control arm.
  Arms: 0g of strawberry

SUMMARY:
The proposed research is designed to extend previous research findings building on the knowledge of strawberries as fruits that support a healthy immune and vascular system. The proposed research leverages a recently funded proposal by the USDA to study in greater depth inflammation, glucoregulation and oxidative stress defense and their relation to improving endothelial function and insulin sensitivity.

Before and after strawberry intake, blood samples will be collected for monocyte (immune cells and source of inflammatory cytokines) isolation and activation via changes in cellular NF-κB and Nrf-2 (key transcription factors of inflammation/oxidative stress defense) status along with products of their activation (ie., plasma cytokines). Because inflammation and oxidative stress impairs endothelial function and insulin sensitivity, acutely and chronically, investigators will also study changes in vascular and insulin sensitivity status, assessing changes in vascular adhesion molecules, endothelial responsiveness through flow mediated vasodilation (ie., FMD) and insulin sensitivity using the Liquid Meal Tolerance (LMTT) if intravenous glucose tolerance test (IVGTT) method cannot be used due to supply chain issues of sterile Dextrose. Glucoregulation will be assessed by placing a Continuous Glucose monitoring (CGM) machine (Dexcom-6) to participants for 10 days at the beginning and at the end of the study period of intervention. The study will be a randomized, double-blinded, 3-arm parallel, 4-week, dose-response study. Individuals with chronic low grade inflammation will be sought to test the anti-inflammation - vaso-relaxing - insulin sensitivity effects of strawberry.

DETAILED DESCRIPTION:
Investigators are proposing to leverage ongoing research funded by USDA to study in greater depth the effect of strawberry intake on chronic low grade inflammation and its relation to endothelial function and insulin sensitivity (InsS). Investigators' rationale is based on facts that inflammation is a key feature in the development of atherosclerotic cardiovascular disease and diabetes, and strawberry intake has been shown to modulate biomarkers of inflammation, but with inconsistencies deserving follow up and better understanding. Of note, meal-induced inflammatory responses seem to be counteracted better with lower amounts of strawberry intake [~1 cup fresh weight equivalent (FWeq) vs 3 cups FWeq]. In contrast, markers of inflammation in the fasting state in humans have been relatively unremarkable showing no or limited change with daily strawberry intake. However, many of these investigations used higher intake levels (~2-3 cup FWeq) to test hypotheses on alternative endpoints (ie., lipids) and in groups with varied health risks. To better understand the effects of strawberry intake on systemic inflammation, investigators propose to study mechanisms (ie., NF-kB/Nrf-2 mediated signaling) within a sub population of immune cells (ie., monocytes) that result in plasma markers of inflammation. Investigators propose to do this by harvesting monocytes from subjects and study the activation of these signaling pathways after 4-week strawberry intake compared to a control condition. To address dose-response dynamics, investigators propose to study two strawberry intake levels (1 cup FWeq and 3 cup FWeq vs Control). Investigators are also interested in expanding recently completed vascular work in our lab showing improved vasodilation (by flow mediated vasodilation) 1 h after strawberry intake and after 4-week strawberry intake (3 cup FWeq) daily in individuals with modestly elevated cholesterol levels. Because chronic inflammation and oxidative stress impair endothelial function, investigators hypothesize that intake levels of strawberry that have the greatest benefit in reducing inflammation and oxidative stress will align with lower markers of endothelial inflammation and enhanced endothelial function (ie., vasodilation). Dietary patterns and components of the diet that preserve or improve endothelial function have an important risk lowering impact on cardiovascular disease development.

And finally, investigators aim to explore more deeply the relationship of strawberry intake, inflammation and InsS using the Liquid Meal Tolerance (LMTT) if intravenous glucose tolerance test (IVGTT) method cannot be used due to supply chain issues of sterile Dextrose. Investigators' previous work with strawberries is suggestive of improved peripheral InsS in a meal-challenge paradigm in overweight individuals with 1 cup FWeq and in abdominally obese individuals and impaired InsS with 3 cup FWeq. Changes in fasting insulin concentrations after intake of strawberries with 1-3 cup FWeq have been neutral.

However, fasting insulin concentrations give insight about liver InsS and less about peripheral InsS, which is relevant in post-meal glucose tolerance. In normal physiology, a major function of insulin in post meal state is to suppress hepatic gluconeogenesis while stimulating glucose uptake into muscle and fat. As impaired InsS is a major risk for developing pre-diabetes and type 2 diabetes, intervening early and strategically with diet, and with specific foods as science supports to restore InsS, is prudent. The proposed research can help characterize the role of strawberries in improving InsS and its relation to inflammation status.

Glucoregulation will be assessed by placing a Continuous Glucose monitoring (CGM) machine (Dexcom-6) which monitors interstitial glucose levels every 5 minutes for 10 days. This will be placed to participants at the beginning of the study for 7-10 days and similarly at the end of the study for 7-10 days of period. The study is focused on three areas important to public health and consumers: inflammation, vascular, and metabolic health. The project will provide new, deeper knowledge in these areas elucidating pathways by which strawberries reduce inflammation and risk for atherosclerotic vascular disease and diabetes. The data can contribute to health claim petitions. The new knowledge can be used to inform/educate a number of stakeholders, including the strawberry industry, consumers, health professionals, the scientific, medical and regulatory communities/agencies, and contribute to the evidence-base for establishing intake recommendations of polyphenolic rich fruits, like strawberries, in the USA, to promote health and reduce chronic disease risk.

ELIGIBILITY:
Inclusion Criteria

* Men or women 20-60 years of age
* High sensitivity C-Reactive Protein (hs-CRP), a global marker of inflammation, >1.0 and ≤10 ng/L
* BMI ≥ 25 kg/m2
* Nonsmokers (Past smokers can be allowed if they have abstinence for minimum of 1 years). Occasional smoker may be allowed at investigator discretion
* Judged to be in good health on the basis of the medical history ie., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, records of food diary and study visit schedule)
* Able to maintain usual physical activity pattern
* Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during study visit

Exclusion Criteria:

* Men and women who smoke regularly
* Men and women with known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at screening visit
* Men and women who have fasting blood glucose concentration >125 mg/dL at screening visit
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc. that, in the opinion of the investigator, could interfere with the interpretation of the study results
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Men and women diagnosed with chronic constipation, diarrhea or other chronic gastrointestinal complaint (e.g. irritable bowel syndrome)
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplement, anti-inflammation, lipid lowering medication, blood pressure lowering medication, etc... Subjects may choose to go off dietary supplements (requires 30-day washout); e.g., fish oil, probiotics, etc...
* Men and women who has participated in prebiotics or laxative trial within 3 months prior to enrollment or any other clinical trial within 1 month
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator.
* Has a known intolerance or sensitivity to any ingredients in the study products
* Has used antibiotics within the previous 2 months
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Unstable weight: gained or lost weight +/- 5 kg (11 lbs) in previous 2 months
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours i.e., working overnight (e.g. 3rd shift)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma biomarkers and measures of inflammation: NF-κB activation/suppression | Baseline to 4 weeks
  The dose related change in measures of inflammation by analyzing NF-κB activation/suppression in monocytes among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).
Change in primary clinical marker of inflammation IL-6 | Baseline to 4 weeks
  The dose related change in blood level of IL-6 among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry). Cellular evaluation of inflammatory status, collected plasma samples will be analyzed for selected inflammatory markers (IL-6) using standard ELISA.

SECONDARY OUTCOMES:
Change flow mediated dilation (FMD) before and after four weeks strawberry intake compared to control | Baseline to 4 weeks
  FMD imaging of the brachial artery is a non-invasive technique that assesses endothelial- dependent relaxation and is used as a surrogate marker of macrovascular endothelial function among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).
Change in Insulin sensitivity index using Liquid Meal Tolerance Test (LMTT). | Baseline to 4 weeks
  Liquid Meal Tolerance Test (LMTT) will be used to assess pre and post intervention fasting insulin sensitivity (HOMA-%S) and rate among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).The IVGTT will be included in a subset only as sterile dextrose is available (supply chain issues).
Change in Beta cell function using Liquid Meal Tolerance Test (LMTT). | Baseline to 4 weeks
  Liquid Meal Tolerance Test (LMTT) will be used to assess pre and post intervention fasting β-cell function (HOMA-%B) and rate among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).The IVGTT will be included in a subset only as sterile dextrose is available (supply chain issues).
Change in Insulin Disposition index using Liquid Meal Tolerance Test (LMTT). | Baseline to 4 weeks
  Liquid Meal Tolerance Test (LMTT) will be used to assess pre and post intervention fasting insulin disposition (HOMA-%S) and rate among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).The IVGTT will be included in a subset only as sterile dextrose is available (supply chain issues).
Change in Insulin Fractional disappearance rate of plasma glucose using Liquid Meal Tolerance Test (LMTT). | Baseline to 4 weeks
  Liquid Meal Tolerance Test (LMTT) will be used to assess pre and post intervention fasting insulin fractional disappearance rate (HOMA-%S) and rate among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).The IVGTT will be included in a subset only as sterile dextrose is available (supply chain issues).
Change in Nrf-2 activation/suppression | Baseline to 4 weeks
  The dose related change in measures of inflammation by analyzing Nrf-2 activation/suppression in monocytes among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).
Change in 10-day Glucose average | Baseline to 4 weeks
  Average glucoregulation will be assessed by using CGM machine (Dexcom-6) by 10 days among participants at the beginning of the intervention and at the end of 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry). This CGM will monitor interstitial glucose levels after placing the machine to participants every 5 minutes for 7-10 days.
Change in fasting Lipids | Baseline to 4 weeks
  The dose related change in measures of fasting Lipids among participants after 4 weeks of strawberry intake (1 cup or 3 cup FWeq) vs control (0 cup strawberry).

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT06173765/ICF_000.pdf